CLINICAL TRIAL: NCT02259296
Title: Timing for Arteriovenous Fistula Creation and Its Effect on Target Organs in Patients With Chronic Renal Failure
Acronym: TACTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Sichuan Provincial People's Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Changlin Mei, Professor, Director, Division of Nephrology, Shanghai Changzheng Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZHKI-HDVA-001
Record Dates: First submitted 2014-09-23; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Renal Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lower eGFR for AVF creation (Experimental)
  Interventions: Procedure: Lower eGFR for AVF construction
- Higher eGFR for AVF creation (Active Comparator)
  Interventions: Procedure: Higher eGFR for AVF construction

INTERVENTIONS:
Procedure: Lower eGFR for AVF construction — Lower eGFR patients (eGFR<10ml/min 1.73m2 for patients without diabetic kidney disease, and eGFR<15ml/min 1.73m2 for diabetic kidney disease) are proposed to undergo AVF construction
  Other Names: late AVF construction
  Arms: Lower eGFR for AVF creation
Procedure: Higher eGFR for AVF construction — Higher eGFR patients (eGFR 10-15ml/min 1.73m2 for patients without diabetic kidney disease, and eGFR 15-20ml/min 1.73m2 for diabetic kidney disease) are proposed to undergo AVF construction
  Other Names: early AVF construction
  Arms: Higher eGFR for AVF creation

SUMMARY:
The timing for arteriovenous fistula (AVF) creation and its effect on target organs in patients with chronic renal failure will be investigated by multicenter prospective cohort. Lower estimated glomerular filtration rate (eGFR) patients (eGFR<10ml/min 1.73m2 for patients without diabetic kidney disease, and eGFR<15ml/min 1.73m2 for diabetic kidney disease) and higher eGFR patients (eGFR 10-15ml/min 1.73m2 for patients without diabetic kidney disease, and eGFR 15-20ml/min 1.73m2 for diabetic kidney disease) will be proposed to undertake AVF creation. Maturation rate and time of AVF will be followed up in 3 months; primary and secondary patency rate of AVF, AVF construction on cardiac structure, function, encephalopathy, cerebral vascular lesions and cognitive function will be followed up in the next 2 years. This multicenter will provide evidence to develop guideline of timing for AVF creation

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal failure, without AVF creation;
* Estimated glomerular filtration rate (eGFR) <15ml/min 1.73m2 for patients without diabetic kidney disease, and eGFR<20ml/min 1.73m2 for diabetic kidney disease;
* All study subjects must agree to participate in the study and provide written informed consent.

Exclusion Criteria:

* Patients with the history of arteriovenous graft, or central venous catheter, or peritoneal dialysis catheter placement;
* Contraindications to AVF construction:

  * Allen's Test is positive, or arterial diameter<2 mm; venous diameter<2.5 mm or venous occlusion/stenosis.
  * Local infection.
* Have any other uncontrolled medical condition (severe heart failure, malignancy, severe coagulation disorders ).
* Mental illness that makes the patients unable to complete the trial.
* Female who is planning to become pregnant, who is pregnant and/or lactating, who is unwilling to use effective means of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Maturation rate of AVF | 3 months
  Assessed by duplex ultrasound. A mature fistula has a flow of over 500 mL/min,is less than 0.6 cm below the surface of the skin, and has a minimal diameter of 0.6 cm
Primary and secondary patency rate of AVF | 2 years
  Assessed by duplex ultrasound

SECONDARY OUTCOMES:
Maturation time of AVF | 3 months
  Assessed by duplex ultrasound
Complications of AVF | 2 years
  Assessed by duplex ultrasound
AVF creation on ventricular volumes and left ventricular remodeling | 2 years
  Assessed by doppler echocardiography
AVF creation on AVF creation on brain MRI and cognitive functions | 2 years
  Cognitive functions are assessed by psychic and autonomy scores

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, Principal Investigator — Division of Nephrology, Changzheng Hospital